CLINICAL TRIAL: NCT04229654
Title: Awareness, Expectations, and Perception of Anomaly Ultrasound Scan Among Pregnant Women in a Northern México Population
Brief Title: Awareness, Expectations, and Perception of Anomaly Scan Among Mexican Pregnant Women
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. med Flavio Hernández Castro, Principal investigator, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: GI15017
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Knowledge; Expectations; Ultrasound
Keywords: knowledge; expectations; anomaly scan
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A written questionnaire was used to capture demographic data, obstetric history, knowledge, expectations, and perception of anomaly scans.

SUMMARY:
To describe the knowledge, expectations, and perception of women towards the mid-trimester ultrasound scan to detect fetal anomalies in a Mexican population.

DETAILED DESCRIPTION:
A cross-sectional survey was conducted in two prenatal diagnostic centers located in Monterrey, Nuevo León, México. One was a university prenatal diagnostic center and the other a private one. The centers were purposively selected to represent different characteristics of the level of care and demographic characteristics. The research instrument was a 26-item questionnaire divided into three sections. The first section contained 12 questions designed to assess women's ideas about the purpose and limitations of the scan (yes/no). The second was on expectations before the scan while the third dealt on women´s perception of the fetus during the ultrasound examination. All women attending for a mid-trimester anomaly scan were invited to fill out the first two parts of a pretested structured questionnaire before the scan and after the ultrasound examination, the third part of the questionnaire concerning their experience of the scan session was completed and collected.

Additionally, the questionnaire included demographic questions (age, parity, educational level, marital status). The source of the questionnaire items was interviews with experts.

Ethical approval for this study was obtained from the Institutional review board. The anomaly scan was performed by fetal-maternal specialists between 18 and 24.6-week gestation.

All data were recorded and analyzed using the Statistical Package for the Social Sciences version 22.0 (SPSS Inc, Illinois, USA). Descriptive statistics were used for the sociodemographic data. Categorical variables were compared using the chi-square test or Fisher exact test. Univariate and multivariate regression analyses were performed to delineate the factors associated with a higher knowledge level. A p-value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

-Pregnant women between 18 and 24.6 weeks

Exclusion Crireria:

* Time constraints
* Lack of interest
* Maternal blindness

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women at 18-24.6 week gestation
Study Population: The study population consisted of pregnant women of gestational age between 18 and 24.6 weeks. Participants were recruited from two prenatal diagnostic centers located in the northern part of México. The centers were purposively selected to represent different characteristics of the level of care and demographic characteristics.
  This study was performed according to the standards of the Helsinki Declaration and approval was obtained from the ethics and educational issues coordinating committee of our University Hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Knowledge | 10 minutes
  Consisted of 12 items that asked about women´s to evaluate the background knowledge about the purpose and limitations of ultrasound anomaly scan. The first three items asked about the women's knowledge and worries about ultrasound and their understanding of the information provided for their attending physicians. The last 3 items were completed after the ultrasound examination, those items asked about opinions regarding the utility and relief of information provided. The correct answers from the other 6 items were summed to form a total score ranging from 0 to 6. The total scores were categorized into three groups: score 0-2 as poor, 3-4 as intermediate, and 5-6 as good.
Expectations | 5 minutes
  Consisted of 8 items that asked about women´s expectations before the ultrasound examination. A yes/no style were used to measure this outcome.
Perception of the fetus | 5 minutes
  Consisted of 6 items that asked about women´s perception of the fetus during ultrasound examination. A yes/no style were used to measure this outcome.

SECONDARY OUTCOMES:
Demographic characteristics | 5 minutes
  Demographic characteristics were collected, including maternal age, body mass index, education level, marital status, gravidity and parity.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Hernández-Castro, MD PhD, Principal Investigator — Universidad Autónoma de Nuevo León
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ugwu AC, Udoh BE, Eze JC, Eze PC. Awareness of information, expectations and experiences among women for obstetric sonography in a south east Nigeria population. East Afr J Public Health. 2011 Jun;8(2):132-4. PMID 22066299
- [Background] Westerneng M, Diepeveen M, Witteveen AB, Westerman MJ, van der Horst HE, van Baar AL, de Jonge A. Experiences of pregnant women with a third trimester routine ultrasound - a qualitative study. BMC Pregnancy Childbirth. 2019 Sep 2;19(1):319. doi: 10.1186/s12884-019-2470-9. PMID 31477046
- [Background] Buyukbayrak EE, Soysal S, Anik Ilhan G, Yavuzer O. What do expectant parents know about antenatal ultrasound screening? J Matern Fetal Neonatal Med. 2020 Jun;33(11):1811-1817. doi: 10.1080/14767058.2018.1530209. Epub 2018 Nov 4. PMID 30261776
- [Background] Bricker L, Garcia J, Henderson J, Mugford M, Neilson J, Roberts T, Martin MA. Ultrasound screening in pregnancy: a systematic review of the clinical effectiveness, cost-effectiveness and women's views. Health Technol Assess. 2000;4(16):i-vi, 1-193. No abstract available. PMID 11070816
- [Background] Garcia J, Bricker L, Henderson J, Martin MA, Mugford M, Nielson J, Roberts T. Women's views of pregnancy ultrasound: a systematic review. Birth. 2002 Dec;29(4):225-50. doi: 10.1046/j.1523-536x.2002.00198.x. PMID 12431263
- [Background] Tautz S, Jahn A, Molokomme I, Gorgen R. Between fear and relief: how rural pregnant women experience foetal ultrasound in a Botswana district hospital. Soc Sci Med. 2000 Mar;50(5):689-701. doi: 10.1016/s0277-9536(99)00321-4. PMID 10658849
- [Background] Salmoukas C, Kundu S, Soergel P, Hillemanns P, von Kaisenberg C, Staboulidou I. Background Knowledge and Attitude of Pregnant Women towards Ultrasound Screening at 20-23 Weeks Gestation. Z Geburtshilfe Neonatol. 2016 Feb;220(1):16-20. doi: 10.1055/s-0035-1545287. Epub 2015 Jun 3. PMID 26039497